CLINICAL TRIAL: NCT02047929
Title: Comparing Traditional and Participatory Dissemination of a Shared Decision Making Intervention
Brief Title: Comparing Types of Implementation of a Shared Decision Making Intervention
Acronym: ADAPT-NC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CD-12-11-4276
Record Dates: First submitted 2014-01-27; First posted 2014-01-28 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Shared decision making; Participatory methods; Practice facilitator; Health coach
MeSH Terms: conditions — Asthma | interventions — SDM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Facilitator-Led (Active Comparator): This approach to dissemination allows clinics some freedom to tailor the Asthma Shared Decision Making (SDM) Toolkit and training process for their specific environment and patient population while maintaining fidelity of certain key elements that are felt to be essential for success. The expertise of the trained Practice Facilitator will help guide the process of implementation at the practice level.
  Interventions: Other: Asthma Shared Decision Making (SDM) Toolkit
- Traditional (Active Comparator): The most commonly used dissemination technique is active diffusion, which includes didactic presentations, academic detailing, exposure to journal publications and subject matter experts, and educational material distribution. We have defined this type of dissemination, "traditional dissemination". For the purpose of this study, practices randomized to traditional dissemination will receive a lunchtime presentation by a physician champion / subject matter expert on shared decision making. The presentation will give an overview of the Asthma Shared Decision Making (SDM) Toolkit, access to the internet link with additional information, and a copy of all printed materials associated with the Toolkit.
  Interventions: Other: Asthma Shared Decision Making (SDM) Toolkit
- Control (No Intervention): A third group will be randomized into an arm with no formal dissemination. This arm will receive information only through passive exposure to the concepts of shared decision making. This would include introduction to the SDM concepts through the media, conferences, or social networks. Having this control in place will allow the research team to isolate the effect of both the FLOW approach and the traditional approach to dissemination.

INTERVENTIONS:
Other: Asthma Shared Decision Making (SDM) Toolkit — A potential solution to improving asthma outcomes is the use of patient-centered approaches like Shared Decision Making (SDM), In the SDM process, patients and their health care providers are engaged jointly in making decisions about medical tests and treatments. The research team for this proposal was funded by the Agency for Health Care Research and Quality to build, disseminate and evaluate a novel Asthma SDM Toolkit - The Asthma Comparative Effectiveness Study. The Toolkit development was completed in 2010 and has been in evaluation for 2 years. This study will continue to evaluate the Toolkit in a wide array of practices across NC while testing a new method of dissemination.
  Arms: Facilitator-Led; Traditional

SUMMARY:
Asthma is a common disease that affects people of all ages and has significant morbidity and mortality. Poor outcomes and health disparities related to asthma result in part from the difficulty of disseminating new evidence and paradigms of care delivery such as shared decision making (SDM) into clinical practice. This study will evaluate a novel mechanism for dissemination of an evidence-based SDM Toolkit for asthma care in primary care practices. The study is ideally suited to study dissemination methods because it will leverage a partnership between an established consortium of practice based research networks (PBRNs) and an advanced Medicaid Network.

This study will evaluate a novel dissemination process (FLOW) to spread an Asthma Shared Decision Making Toolkit to practices within a Medicaid network using a consortium of practice-based research networks (NCNC). The knowledge gained from this proposal and the partnerships formed between practice-based research networks and NC Medicaid will facilitate widespread dissemination to almost 300 practices.

DETAILED DESCRIPTION:
Changing the behavior of health providers can be challenging, and significant gaps exist in our knowledge of how to best disseminate new medical evidence into everyday practice. This is true when the evidence involves a new paradigm of patient-centered care delivery such as shared decision making (SDM). The most common dissemination used is passive diffusion, which includes journal publications, didactic presentations, and educational material and often fails to produce timely or sustainable practice level changes. A unique partnership between a Medicaid network and a well established consortium of practice-based research networks provides an ideal venue to examine the effectiveness of new effective methods of dissemination. We previously developed an asthma toolkit that was funded by the Agency for Healthcare Research and Quality (AHRQ) and tested across a regional network of Pediatric, Family Medicine, and Internal Medicine ambulatory practices in Mecklenburg County North Carolina. During this study, key principles of community based participatory research were used engaging providers and patients to develop a Facilitator-Led participant OWned (FLOW) Approach to dissemination. The FLOW approach uses Practice Facilitators to guide practices through the process of adapting the Toolkit into the existing culture and workflow. This approach led to rapid dissemination and sustainability of the Toolkit across six practices. The initial results have showed marked improvement in patient outcomes (improved medication adherence and decreased asthma exacerbations) with increased patient involvement in the creation of the care plans. The objective is to determine what dissemination strategy most effectively increases practice level adoption of shared decision making, improves patient outcomes, and increases patient involvement in care decisions. We will leverage a partnership between the statewide Medicaid network and NCNC, a state-wide consortium of research networks, to identify best practices for dissemination of the shared decision making toolkit. We will test the FLOW method for dissemination on a larger scale by randomizing 30 primary care practices from 4 practice based research networks to one of three dissemination arms: (1) Facilitator-Led participant OWned (FLOW) Approach to Dissemination; (2) Traditional dissemination (Active Diffusion) with facilitator exposure; and (3) Passive dissemination.

ELIGIBILITY:
Inclusion Criteria: North Carolina practices will be eligible for participation in the study if they have over 75 active Medicaid patients in their panel with the diagnosis of asthma.

-

Exclusion Criteria: Prior participation in the Asthma Comparative Effectiveness Study.

-

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Tapp, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Department of Family Medicine, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Shade L, Reeves K, Rees J, Hendrickson L, Halladay J, Dolor RJ, Bray P, Tapp H. Research nurses as practice facilitators to disseminate an asthma shared decision making intervention. BMC Nurs. 2020 May 18;19:40. doi: 10.1186/s12912-020-00414-0. eCollection 2020. PMID 32477003
- [Derived] Ludden T, Shade L, Welch M, Halladay J, Donahue KE, Coyne-Beasley T, Bray P, Tapp H. What types of dissemination of information occurred between researchers, providers and clinical staff while implementing an asthma shared decision-making intervention: a directed content analysis. BMJ Open. 2020 Mar 8;10(3):e030883. doi: 10.1136/bmjopen-2019-030883. PMID 32152153
- [Derived] Shade L, Ludden T, Dolor RJ, Halladay J, Reeves K, Rees J, Hendrickson L, Bray P, Tapp H. Using the Consolidated Framework for Implementation Research (CFIR) to evaluate implementation effectiveness of a facilitated approach to an asthma shared decision making intervention. J Asthma. 2021 Apr;58(4):554-563. doi: 10.1080/02770903.2019.1702200. Epub 2019 Dec 23. PMID 31868043
- [Derived] Tapp H, McWilliams A, Ludden T, Kuhn L, Taylor Y, Alkhazraji T, Halladay J, Derkowski D, Mohanan S, Dulin M. Comparing traditional and participatory dissemination of a shared decision making intervention (ADAPT-NC): a cluster randomized trial. Implement Sci. 2014 Oct 29;9:158. doi: 10.1186/s13012-014-0158-0. PMID 25359128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All practices were recruited and randomized by May 2014.
Pre-assignment Details: All practices were randomized in the study. Since the intervention was practice wide, individual patients were not required to be enrolled or consented.
Units Other Than Participants: Primary Care Practices
Groups:
- Facilitator-Led Participant Owned (FLOW) Dissemination: This approach to dissemination allows clinics some freedom to tailor the SDM Toolkit and training process for their specific environment and patient population while maintaining fidelity of certain key elements that are felt to be essential for success. The expertise of the trained Practice Facilitator will help guide the process of implementation at the practice level.
  Asthma Shared Decision Making (SDM) Toolkit: A potential solution to improving asthma outcomes is the use of patient-centered approaches like Shared Decision Making (SDM), identified by both the Institute of Medicine and the Patient-Centered Outcomes Research Institute as an important new means of improving patient outcomes. In the SDM process, patients and their health care providers are engaged jointly in making decisions about medical tests and treatments. This study will continue to evaluate the Toolkit in a wide array of practices across NC while testing a new method of dissemination.
- Traditional Dissemination (Active Diffusion): The most commonly used dissemination technique is active diffusion, which includes didactic presentations, academic detailing, exposure to journal publications and subject matter experts, and educational material distribution. We have defined this type of dissemination, "traditional dissemination". For the purpose of this study, practices randomized to traditional dissemination will receive a lunchtime presentation by a physician champion / subject matter expert on shared decision making. The presentation will give an overview of the Asthma SDM Toolkit, access to the internet link with additional information, and a copy of all printed materials associated with the Toolkit.
Period: Overall Study
Arm/Group | Facilitator-Led Participant Owned (FLOW) Dissemination | Traditional Dissemination (Active Diffusion) | Control
Started | 1503; 10 Primary Care Practices | 2523; 10 Primary Care Practices | 2248; 10 Primary Care Practices
Practice Rollout | 1503; 10 Primary Care Practices | 2523; 10 Primary Care Practices | 0; 0 Primary Care Practices (Per protocol, practice did not receive any intervention from practice facilitator)
Practice Refresher | 1503; 10 Primary Care Practices | 2523; 10 Primary Care Practices | 0; 0 Primary Care Practices (Per protocol, practices did not receive any interaction from practice facilitator)
Surveys Collected | 1503; 10 Primary Care Practices | 2523; 10 Primary Care Practices | 0; 0 Primary Care Practices (Per protocol, practice did not receive any interaction from practice facilitator)
Completed | 1503; 10 Primary Care Practices | 2523; 10 Primary Care Practices | 2248; 10 Primary Care Practices
Not Completed | 0; 0 Primary Care Practices | 0; 0 Primary Care Practices | 0; 0 Primary Care Practices

BASELINE CHARACTERISTICS:
Population: Number of Medicaid patients diagnosed with Asthma
Groups:
- Total: Total of all reporting groups
Arm/Group | Facilitator-Led Participant Owned (FLOW) Dissemination | Traditional Dissemination (Active Diffusion) | Control | Total
Number analyzed (Participants) | 1503 | 2523 | 2248 | 6274
Age, Customized [Count of Participants; unit: Participants]
  Under the Age of 21 | 1340 | 2223 | 2058 | 5621
  Age 21 and Older | 163 | 300 | 190 | 653
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 670 | 1121 | 950 | 2741
  Male | 833 | 1402 | 1298 | 3533

OUTCOME MEASURES:

1. Primary Outcome: Patient Perception of Shared Decision Making
Description: Success of the dissemination process will be determined by looking at process and outcome measures collected at the patient and clinic level. The primary outcome will be the patient's perceptions of shared decision making using a patient survey.
Time Frame: 18 months
Population: Number of surveys collected. Per the protocol, surveys were not collected for the Usual Care cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Facilitator-Led: This approach to dissemination allows clinics some freedom to tailor the Asthma Shared Decision Making (SDM) Toolkit and training process for their specific environment and patient population while maintaining fidelity of certain key elements that are felt to be essential for success. The expertise of the trained Practice Facilitator will help guide the process of implementation at the practice level.
  Asthma Shared Decision Making (SDM) Toolkit: A potential solution to improving asthma outcomes is the use of patient-centered approaches like Shared Decision Making (SDM), In the SDM process, patients and their health care providers are engaged jointly in making decisions about medical tests and treatments. The research team for this proposal was funded by the Agency for Health Care Research and Quality to build, disseminate and evaluate a novel Asthma SDM Toolkit - The Asthma Comparative Effectiveness Study. The Toolkit development was completed in 2010 and has been in evaluation for
- Traditional: For the purpose of this study, practices randomized to traditional dissemination will receive a lunchtime presentation by a physician champion / subject matter expert on shared decision making. The presentation will give an overview of the Asthma Shared Decision Making (SDM) Toolkit, access to the internet link with additional information, and a copy of all printed materials associated with the Toolkit.
  Asthma Shared Decision Making (SDM) Toolkit: A potential solution to improving asthma outcomes is the use of patient-centered approaches like Shared Decision Making (SDM), In the SDM process, patients and their health care providers are engaged jointly in making decisions about medical te
Arm/Group | Facilitator-Led | Traditional
Number analyzed (Participants) | 705 | 523
Participants
  The provider alone made the decision | 34 | 40
  The provider mostly made the decision, and I playe | 86 | 79
  The provider and I participated equally in making | 528 | 347
  I mostly made the decision, and the provider play | 30 | 26
  I alone made the decision | 27 | 31

2. Secondary Outcome: Health Outcomes
Description: Health outcomes data collected from Continuing Care of North Carolina that indicate poor asthma control and/or marker for exacerbations. These include patients with: Emergency Department Visits, Hospitalizations, Oral Steroid prescriptions, or patients with one or more of the markers for exacerbation: Emergency Department Visits, Hospitalizations, Oral Steroid prescriptions.
Time Frame: 18 months
Population: Medicaid Patients diagnosed with Asthma
Measure: Count of Participants; unit: Participants
Arm/Group | Facilitator-Led Participant Owned (FLOW) Dissemination | Traditional Dissemination (Active Diffusion) | Control
Number analyzed (Participants) | 1503 | 2523 | 2248
Participants
  Patients with Emergency Department Visits | 144 | 355 | 288
  Patients with Hospitalizations | 23 | 29 | 38
  Patients with Oral Steroid Prescriptions | 550 | 977 | 764
  Patients with Exacerbations | 599 | 1031 | 810

3. Secondary Outcome: Medication Adherence
Description: Additional measures that will be evaluated to determine the success of dissemination will be based on indicators of poor asthma control including: medication adherence (controller medication refills). Data was not collected.
Time Frame: 18 months
Population: Data was not collected
Groups:
- Traditional: We have defined this type of dissemination, "traditional dissemination". For the purpose of this study, practices randomized to traditional dissemination will receive a lunchtime presentation by a physician champion / subject matter expert on shared decision making. The presentation will give an overview of the Asthma Shared Decision Making (SDM) Toolkit, access to the internet link with additional information, and a copy of all printed materials associated with the Toolkit.
  Asthma Shared Decision Making (SDM) Toolkit: A potential solution to improving asthma outcomes is the use of patient-centered approaches like Shared Decision Making (SDM), In the SDM process, patients and their health care providers are engaged jointly in making decisions about medical te
Arm/Group | Facilitator-Led | Traditional | Control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Data was not collected as part of this trial. Intervention was applied to the whole clinic and individual patients were not tracked by the research team. Survey data was anonymous and occurred right after clinic visit. Outcomes data collected for this project came through summarized data provided by the state Medicaid network where adverse events are not collected.
Description: Adverse Event Data was not collected as part of this trial. Intervention was applied to the whole clinic and individual patients were not tracked by the research team. Survey data was anonymous and occurred right after clinic visit. Outcomes data collected for this project came through summarized data provided by the state Medicaid network where adverse events are not collected.
Arm/Group | Facilitator-Led Participant Owned (FLOW) Dissemination | Traditional Dissemination (Active Diffusion) | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to system data changes with our secondary outcomes data source, medication adherence was not collected for the study. Age data was only collected based under the age of 21 and 21 and older.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes